CLINICAL TRIAL: NCT06906510
Title: Evaluation of Trimethylamine N-oxide (TMAO) Levels in Periodontal Disease
Acronym: TMAO
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Collaborators: Istanbul Medipol University Hospital (Other); Ankara University (Other); Acibadem University (Other); Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Ceyhan CERAN SERDAR, Assistant Prof., Ankara Medipol University
Other Study IDs: 1004
Record Dates: First submitted 2025-03-13; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Inflammation; Trimethylamine N-oxide (TMAO); TNF-alfa
Keywords: periodontal disease; TMAO; TNF-α; periodontitis
MeSH Terms: conditions — Periodontitis; Inflammation; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Individuals: Systemically healthy individuals without periodontitis
  Interventions: Diagnostic Test: Salivary and Serum TMAO Mesurement; Diagnostic Test: Salivary and Serum TNF-α Mesurement
- Patients with Periodontitis: Systemically healthy individuals with periodontitis
  Interventions: Diagnostic Test: Salivary and Serum TMAO Mesurement; Diagnostic Test: Salivary and Serum TNF-α Mesurement

INTERVENTIONS:
Diagnostic Test: Salivary and Serum TMAO Mesurement — Salivary and serum TMAO levels were measured by liquid chromatography-mass spectrometry (LC-MS/MS)
Diagnostic Test: Salivary and Serum TNF-α Mesurement — Salivary and serum TNF-α levels were measured by ELISA

SUMMARY:
Salivary and serum levels of TMAO and TNF-α can distinguish between individuals with periodontitis and periodontally healthy individuals.

DETAILED DESCRIPTION:
Trimethylamine N-oxide (TMAO), a gut flora-derived metabolite from dietary choline, has emerged as an indicator of atherosclerosis. Circulatory TMAO has been implicated in cardiovascular risks by altering enterohepatic cholesterol and bile acid metabolism, increasing macrophage scavenger receptor expression, and activating nuclear factor kappa B (NF-κB) via pro-inflammatory genes such as interleukin-1 (IL-1). The pro-inflammatory cytokine tumor necrosis factor-alpha (TNF-α), which plays a crucial role in immune responses and inflammation, has been demonstrated as a crucial participant also during the development of periodontal diseases. The aim of this study is to evaluate difference in salivary and serum levels of TMAO and TNF-α between individuals with periodontitis and periodontally healthy individuals.

The study includes two groups: systemically and periodontally healthy control subjects (n= 24), and patients with periodontitis (n=24). Periodontal parameters were recorded. TMAO levels in saliva and serum were determined by liquid chromatography-mass spectrometry (LC-MS/MS), and TNF-α levels were determined by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 and under 65 years of age;
* having at least 20 natural teeth excluding the third molars; and
* being systemically healthy.

Exclusion Criteria:

* being smoker;
* chronic use of any systemic medication
* use of antibiotics and/or anti-inflammatory steroids, nonsteroidal anti-inflammatory drugs, immunosuppressants, beta-blockers, calcium channel blockers, anticoagulants, or hormonal contraceptives within 3 months preceding the study;
* pregnancy or lactation; and
* use of orthodontic appliances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy individuals who applied to the Department of Periodontology at Istanbul Medipol University, Faculty of Dentistry between January 2024 and August 2024.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) | Baseline
  Clinical parameters such as Probing depth (PD), Plaque index (PI), Bleeding on probing (BOP), and Clinical attachment loss (CAL) were recorded.
Plaque index (PI) | Baseline
  Clinical parameters such as Probing depth (PD), Plaque index (PI), Bleeding on probing (BOP), and Clinical attachment loss (CAL) were recorded.
Bleeding on probing (BOP) | Baseline
  Clinical parameters such as Probing depth (PD), Plaque index (PI), Bleeding on probing (BOP), and Clinical attachment loss (CAL) were recorded.
Clinical attachment loss (CAL) | Baseline
  Clinical parameters such as Probing depth (PD), Plaque index (PI), Bleeding on probing (BOP), and Clinical attachment loss (CAL) were recorded.
Age | Baseline

SECONDARY OUTCOMES:
Salivary and serum TMAO | Baseline
  Salivary and serum TMAO and TNF-α levels are measured.
  Participants were instructed to rinse their mouths using filtered water and seated calmly while they spit into a disposable tube for five minutes, and saliva was collected from all patients. Saliva samples were prepared for storage by centrifugation at 3000 ×g for 10 minutes.
  Standard venipunctures were used to collect blood; the samples were stored at room temperature for 30 minutes. Serum was prepared from blood samples by centrifugation at 4000 ×g for 10 minutes.
  All serum and saliva samples have been transferred into Eppendorf tubes and preserved at -80oC until the analysis date.
  Salivary and serum TMAO levels were analyzed by LC-MS/MS. Salivary and serum TNF-α levels were measured using a commercial ELISA kit.
Salivary and serum TNF-α levels | Baseline
  Salivary and serum TMAO and TNF-α levels are measured.
  Participants were instructed to rinse their mouths using filtered water and seated calmly while they spit into a disposable tube for five minutes, and saliva was collected from all patients. Saliva samples were prepared for storage by centrifugation at 3000 ×g for 10 minutes.
  Standard venipunctures were used to collect blood; the samples were stored at room temperature for 30 minutes. Serum was prepared from blood samples by centrifugation at 4000 ×g for 10 minutes.
  All serum and saliva samples have been transferred into Eppendorf tubes and preserved at -80oC until the analysis date.
  Salivary and serum TMAO levels were analyzed by LC-MS/MS. Salivary and serum TNF-α levels were measured using a commercial ELISA kit.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khanna S, Mali AM. Evaluation of tumor necrosis factor-alpha (TNF-alpha) levels in plasma and their correlation with periodontal status in obese and non-obese subjects. J Indian Soc Periodontol. 2010 Oct;14(4):217-21. doi: 10.4103/0972-124X.76920. PMID 21731245
- [Background] Engebretson S, Chertog R, Nichols A, Hey-Hadavi J, Celenti R, Grbic J. Plasma levels of tumour necrosis factor-alpha in patients with chronic periodontitis and type 2 diabetes. J Clin Periodontol. 2007 Jan;34(1):18-24. doi: 10.1111/j.1600-051X.2006.01017.x. Epub 2006 Nov 20. PMID 17116158
- [Background] Buczko P, Zalewska A, Szarmach I. Saliva and oxidative stress in oral cavity and in some systemic disorders. J Physiol Pharmacol. 2015 Feb;66(1):3-9. PMID 25716960
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Hernandez-Ruiz P, Escalona Montano AR, Amezcua-Guerra LM, Gonzalez-Pacheco H, Niccolai E, Amedei A, Aguirre-Garcia MM. Potential Association of the Oral Microbiome with Trimethylamine N-Oxide Quantification in Mexican Patients with Myocardial Infarction. Mediators Inflamm. 2024 Feb 20;2024:3985731. doi: 10.1155/2024/3985731. eCollection 2024. PMID 38415052
- [Background] Zhou J, Chen S, Ren J, Zou H, Liu Y, Chen Y, Qiu Y, Zhuang W, Tao J, Yang J. Association of enhanced circulating trimethylamine N-oxide with vascular endothelial dysfunction in periodontitis patients. J Periodontol. 2022 May;93(5):770-779. doi: 10.1002/JPER.21-0159. Epub 2021 Nov 3. PMID 34472093
- [Background] Yang T, Santisteban MM, Rodriguez V, Li E, Ahmari N, Carvajal JM, Zadeh M, Gong M, Qi Y, Zubcevic J, Sahay B, Pepine CJ, Raizada MK, Mohamadzadeh M. Gut dysbiosis is linked to hypertension. Hypertension. 2015 Jun;65(6):1331-40. doi: 10.1161/HYPERTENSIONAHA.115.05315. Epub 2015 Apr 13. PMID 25870193
- [Background] Wu K, Yuan Y, Yu H, Dai X, Wang S, Sun Z, Wang F, Fei H, Lin Q, Jiang H, Chen T. The gut microbial metabolite trimethylamine N-oxide aggravates GVHD by inducing M1 macrophage polarization in mice. Blood. 2020 Jul 23;136(4):501-515. doi: 10.1182/blood.2019003990. PMID 32291445